CLINICAL TRIAL: NCT05631275
Title: The Role of Bioimpedance Analysis in Diagnosis and Evaluation of Patients With Chronic Heart Failure and Systolic Ventricular Dysfunction. Correlation of This Tool With Other Heart Failure Markers
Brief Title: The Role of Bioimpedance Analysis in Patients With Chronic Heart Failure and Systolic Ventricular Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Rocio Carda Barrio, MhD, PhD, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Other Study IDs: PIC003-20_FJD
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure (HF) represents a major problem in today's health care landscape and is expected to grow in the next years due to an aging population and improved treatments. In many cases, the evaluation of the volemia status of patients with left ventricular dysfunction is not easy in the outpatient setting, due to limitations of physical examination in stable patients, as well as the tolerance to chronic HF they have. The aim of this study is to determine whether the bioelectrical impedance analysis (BIA) is useful in determining the real clinical stability of chronic HF, its potential implications for clinical management and patient follow-up, as well as for the adjustment of pharmacological treatment. This study is observational, single-center, single-blind and outpatient. It includes patients with a previous diagnosis of HF and left ventricular ejection fraction (LVEF) ≤ 40%, who are stable at the time of inclusion. Follow-up is estimated to be 12 months.

DETAILED DESCRIPTION:
Endpoints:

The primary end-point is to determine the volemia status of the patients and whether there is a correlation between clinical and analytical parameters and those determined with the BIA. It will also be correlated with the clinical questionnaire (ICEBERG). Secondary objectives: to analyze whether the data obtained with BIA correlate with heart failure events such as hospitalization, change in the functional class of patients, worsening renal function, need for changes in medical treatment or implantation of intracardiac devices. In addition, if data allows it, we will evaluate the relationship with quality of life, cardiovascular mortality, changes in biomarkers (NT-ProBNP (N-terminal pro-B-type natriuretic peptide), Troponin I...), and cost-effectiveness.

Design:

This study was design as a single-center observational study in which patients undergoing to a cardiology consultation were selected and underwent bioimpedance measurement as well as a clinical questionnaire. The aim is to obtain data that will help the execution of a larger study about a broadly use of BIA in the management of HF in the future. This study was approved by an institutional review committee and performed under Helsinki Declaration Guidelines. All patients signed the informed consent before entering the study.

The study population is outpatients attended at cardiology consultations of the Hospital Universitario Fundación Jiménez Díaz, with a diagnosis of stable HF (without admission due to decompensation or first episode of HF in the previous year) and with a LVEF ≤ 40% will be included. We estimate that approximately 100 patients can be included in a 3-month inclusion period.

Study procedures: The variables collected are general medical data, analytical data, including the cardiac biomarker NT-proBNP and answers to the ICEBERG questionnaire. BIA is performed when the patient is included in the study.

For follow-up, a review of the clinical history will be carried out in the next months, including a phone contact with the patient if necessary, to obtain information related to mortality or hospital care due to chronic HF.

ELIGIBILITY:
Inclusion Criteria:

- Outpatients attended at cardiology consultations of the Hospital Universitario Fundación Jiménez Díaz, with a diagnosis of stable HF and with a LVEF ≤ 40%.

Exclusion Criteria:

* admission due to decompensation or first episode of HF in the previous year
* amputated patients
* Chronic treatment with corticosteroids
* Pregnancy and breastfeeding
* Any clinically significant condition detected at the time of screening that in the opinion of the investigators may impair the safe completion of the study or limit the evaluation of the endpoints.
* Patients who are actively participating in clinical trials other than observational trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is outpatients attended at cardiology consultations of the Hospital Universitario Fundación Jiménez Díaz, with a diagnosis of stable HF (without admission due to decompensation or first episode of HF in the previous year) and with a LVEF ≤ 40%
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2023-09-07 (Estimated)

PRIMARY OUTCOMES:
Patients Volemia status | 15 minutes
  determine the volemia status of the patients with the BIA parameters

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gaebelt, MD, PhD, Study Director — Fundación Jiménez Dia University Hospital, IIS-FJD
Locations (1):
- Fundación Jiménez Dia University Hospital, IIS-FJD, Madrid, Spain